CLINICAL TRIAL: NCT06015581
Title: Scaling Up Implementation Strategies to Improve the DIAGNOSE and PREVENT Pillars for Young MSM in Florida
Acronym: YACHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: University of Pennsylvania (Other); Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00003373
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped Wedged Design with a second randomization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Implementation Package (Experimental): Continuous Quality Improvement (CQI)
  Interventions: Behavioral: Workforce Development: Tailored Motivational Interviewing and Technical Assistance; Behavioral: Quality Management, Mystery Shopper Feedback
- Observation (Other): Usual Care
  Interventions: Behavioral: Quality Management, Mystery Shopper Feedback
- EPIS Qualitative (No Intervention): 5 providers of 42 sites will participate in Exploration, Preparation, Implementation, Sustainment (EPIS) qualitative interviews (N=210)

INTERVENTIONS:
Behavioral: Workforce Development: Tailored Motivational Interviewing and Technical Assistance — TMI training includes an initial 12 hour virtual workshop, standard patient interaction with feedback, group coaching, and a final standard patient interaction and feedback. TMI relies on experiential activities developed by the network while minimizing didactic presentations. Stigma-reducing communication is emphasized by practicing autonomy supportive and empathic statements and improving cultural humility practices. Role plays map on to the Mystery Shopper domains focusing on risk reduction counseling and PrEP referral. TA addresses factors in the EPIS framework.
  Arms: Implementation Package
Behavioral: Quality Management, Mystery Shopper Feedback — Mystery shoppers visit each agency two times per quarter to systematically examine testing clinics' environmental characteristics and their experiences with clinic staff (e.g., quality of testing session, safer sex discussions, perceived provider competency, PrEP discussions and referral). The investigator team meets with each agency once per quarter to review the data and provide technical assistance.
  Arms: Implementation Package; Observation

SUMMARY:
In this study, investigators will test the YACHT package in 42 FDOH contracted Counseling, Testing and Referral (CTR) agencies across Florida's seven End the HIV Epidemic (EHE) counties. The study is powered on both effectiveness outcomes (number of HIV tests of Young Sexual Minority Men - YSMM) and implementation outcomes, consistent with a type 2 hybrid trial. It is hypothesized that YACHT will improve providers' fidelity to Tailored Motivational Interviewing (TMI) when delivering risk reduction counseling (RRC) and PrEP referrals (implementation outcomes) and will increase testing among YSMM (effectiveness outcome). Investigators will use an innovative stepped wedge design to test the YACHT package, including a second randomization to explore ongoing quality management (QM) with mystery shoppers (MS) as a sustainment strategy. The study also contains a qualitative component based on the Exploration, Preparation, Implementation, Sustainment (EPIS) framework to further understand the context of implementation and sustainment (sequential explanatory mixed methods).

DETAILED DESCRIPTION:
Primary Aim: To test the effect of YACHT to improve fidelity to DIAGNOSE and PREVENT EBPs in 42 FDOH contracted CTR agencies in the seven Florida EHE counties. The primary effectiveness outcome is the number of HIV tests among YSMM. The primary implementation outcome is developmentally and culturally responsive delivery of competent EBPs (RRC, PrEP referral, TMI) based on MS assessments.

Secondary Aim 1: To assess the effect of continued QM (ongoing MS feedback) in sustaining the primary outcomes.

Secondary Aim 2: To utilize mixed methods based on the EPIS framework to understand barriers and facilitators of successful implementation and sustainment of youth-specific EBPs within CTR to improve the DIAGNOSE and PREVENT pillars for YSMM.

In the proposed study, investigators will test the YACHT package in 42 FDOH contracted CTR agencies across Florida's seven EHE counties. The study is powered on both effectiveness outcomes (number of HIV tests of YSMM) and implementation outcomes (EBP fidelity), consistent with a type 2 hybrid trial. The investigative team hypothesizes that YACHT will improve providers' fidelity to TMI when delivering RRC and PrEP referrals (implementation outcomes) and will increase testing among YSMM (effectiveness outcome). The study will use an innovative stepped wedge design to test the YACHT package, including a second randomization to explore ongoing QM with MS as a sustainment strategy.

Primary effectiveness outcome: The primary outcome is # of tests of YSMM (ages 15-29), as reported in aggregate at the agency- and county-level. Investigators expect that the YACHT package will improve the number of HIV tests administered to YSMM at each agency. As an exploratory outcome, FDOH has recently begun tracking PrEP uptake, defined as ≥1 day of TDF/FTC prescribed for PrEP. Both the testing and PrEP data are currently reported in a standardized fashion to FDOH. Data will be aggregated within agencies and will be requested biannually. Data will be managed into quarterly windows to correspond to the data collection intervals in the stepped wedge design.

Primary implementation outcomes: Procedures for MS are described in C4a Exploration and domains are described in Preliminary Studies (section C1c). Using the pre-established MS domains, investigators will compute an overall agency score using the pooled scores from the two MS conducted each quarter. Pooled scores will be presented to reduce potential selection bias and confounding based on whether the same or a different provider interacted with the shoppers at either agency visit, and to account for the variability across shoppers. Domain sub-scores will also be created using psychometrically tested subscales for: 1) LGBT visibility, 2) medical form inclusivity, 3) perceived clinic environment, 4) privacy and confidentiality, 5) relationship context, 6) RRC, 7) safer sex education, 8) PrEP information and referral, 9) perceived provider competency, and 10) patient-provider interactions. For ease of interpretability across domains, investigators will normalize the pooled average scores into percentiles.

ELIGIBILITY:
Inclusion Criteria:

* Site inclusion: All Florida Department of Health (FDOH) contracted or direct service agencies (k=42) across all seven EHE counties that meet eligibility criteria: 1) provide HIV CTR, and 2) tested a minimum of 24 tests to YSMM in the last year.
* Provider Inclusion: Provide CTR at eligible sites.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2027-05-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Testing of YSMM from FDOH Surveillance | 54 months plus 12 months prior to the study start
  The outcomes will be the count of HIV tests delivered to YSMM
Service quality via Mystery Shopper Assessments composite | Quarterly from Month 7 to Month 54
  Two mystery shoppers visit each agency once per quarter. Using the pre-established MS domains (Session Speed, LGBT Visibility, Medical Forms, Clinic Environment, Privacy and Confidentiality, PrEP-specific Indicators, Relationship Context, Counseling Session, Safer Sex Education, Perceived Provoder Competency, Provider Interactions), we will compute an overall agency score using the pooled scores from the two MS conducted each quarter.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Center for Translational Behavioral Science, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Giguere R, Fernandez MI, Bauermeister JA, Balan IC, Aryal S, Cheshure A, Green S, Lin W, Morgan J, Naar S. The Young Adult Centered Healthforce Training (YACHT) Program to Increase HIV Testing and Pre-Exposure Prophylaxis Referrals Among Young Sexual Minority Men in Florida: Protocol for a Type 2 Implementation-Effectiveness Hybrid Trial With a Stepped Wedge Design. JMIR Res Protoc. 2024 Nov 20;13:e63191. doi: 10.2196/63191. PMID 39566048